CLINICAL TRIAL: NCT04482010
Title: Sanu Gundo (jòli sègèsègèli - furakèli - jàntoli): Survey on the Feasibility of the Community-based HIV Care, and Its Impact on Access and Retention in Care in Artisanal Gold Mining Zones in Mali
Brief Title: ANRS 12392 Sanu Gundo
Acronym: SANU GUNDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: UMR 1252 SESSTIM (Unknown); ARCAD Santé PLUS (Unknown); SEREFO (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ANRS 12392
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections
Keywords: Linkage-to-care and retention; Community-based research; Informal gold mining zones; Mali
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: ARCAD Santé PLUS NGO will offer community-based activities of HIV prevention and screening during 5 months. 8833 people will be tested for HIV in the two artisanal gold-mining sites. Thus, 265 HIV-positive individuals will be enrolled:
  * Control group: 129 (Diassa), 30% of attrition and 5% of discordant HIV screening and confirmatory tests;
  * Intervention group: 136 (Kofoulatiè), 30% of attrition; 5% of people accepting the study but refusing the community-based HIV care; and 5% of discordant HIV screening and enrolment tests.
  This is the minimum number required to verify the primary endpoint of the study. The intervention consists in the provision of community-based healthcare services for HIV provided by ARCAD Santé PLUS's members in the Kofoulatiè site. People in the Diassa site (control group) will be referred to the public healthcare centers for classic HIV care. A quantitative survey with follow-up at M1, M3, M6, M9 and M12 after HIV diagnosis.
Who Masked: Participant
Masking Description: Participants in the control group (HIV positive people at the artisanal gold-mining site in Diassa) will not be aware of the existence of the community-based HIV care services provided by ARCAD Santé PLUS at the Kofoulatiè artisanal gold-mining site.
  The distance between these sites is around 400km. However they share similar characteristics in terms of geographical localisation, size and healthcare supply.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic HIV care (No Intervention): Participants diangosed HIV positive at the time of the community-based activities conducted by ARCAD Santé PLUS. They will be referred to the referral centers (CSRéf) for the classic HIV care in the Malian public health system.
- Community-based HIV care (Other): Participants diagnosed HIV positive at the time of the community-based activities by ARCAD Santé PLUS. They will receive community-based HIV care by the NGO at the gold-mining site.
  Interventions: Other: Local community-based HIV care

INTERVENTIONS:
Other: Local community-based HIV care — Compared to the classic HIV care, community-based HIV care includes:
  * Individual interviews with a psychosocial agent;
  * Support groups conducted by psychosocial agents;
  * Culinary workshops gathering PLWHIV and healthcare professionals;
  * Home visits by a community worker;
  * Emergency relief based on a funding for patients with urgent needs
  As in the classic HIV care, ARCAD Santé PLUS provides consultations with doctors, prescriptions and delivery of antiretroviral (ARV) treatment every 3 months, biological analyses for enrolment, and follow-up every 6 months. In addition, psychosocial agents from ARCAD Santé PLUS propose workshops on education and support for adherence to treatment.
  Arms: Community-based HIV care

SUMMARY:
Sanu Gundo ANRS 12392 is a non-randomized and non-comparative intervention trial in Mali.

The main objective of the project is to study the feasibility of the community-based HIV care in the context of the artisanal gold mining zones and to evaluate its contribution to the linkage-to-care of PLWHIV with the health system and their retention in care, as well as its effect on their health status.

DETAILED DESCRIPTION:
Convergence of key-populations in the informal gold mining zones suggests the important exposure to HIV contamination of people living in these zones. The pilot project Sanu Gundo showed a prevalence of 8% in the site of Kokoyo, much higher than the 1.1% national prevalence. The large rates of HIV patients lost to followup underline the difficulties experienced by the health system. Introducing a community-based HIV care offer in proximity to people in the informal gold mining zones could contribute to the improvement not only of access to HIV prevention and testing, but also to the access and retention in care.

Sanu Gundo ANRS 12392 is a non-randomized and non-comparative intervention trial. Community-based activities conducted by ARCAD Santé PLUS (during 5 months) including HIV testing will contribute to the construction of both a control and intervention groups. These groups will be formed by people tested positive to HIV during the community-based activities conducted by ARCAD Santé PLUS in two artisanal gold mining sites.

The control group will include 129 participants positive to HIV in Diassa (Sikasso region), and the intervention group will include 136 participants positive to HIV in Kofoulatiè (Koulikoro region).

The intervention consists local community-based activities for HIV care provided by ARCAD Santé PLUS for people living in Kofoulatiè (intervention group), whereas people living in Diassa (control group) will be referred to the Referral Health Centers (CSRéf) as recommended by the national guidelines.

The total number of 265 participants diagnosed positive to HIV enrolled in the study corresponds (at least) to the HIV prevalence of 3% observed during the first two months of participants enrolment (November 2020 to January 2021). Accounting for survey attrition, refusal of the community-based HIV care and non-inclusion criteria, it is expected that 172 participants (86 per group) will be followed-up during the whole duration of the study. This corresponds to the number of participants required to verify the primary endpoint of the study: a better retention rate in healthcare 12 months after of HIV diagnosis for people receiving community-based care by ARCAD Santé PLUS.

A quantitative survey will be conducted with the administration of questionnaires at different point-times during the follow-up for HIV care: M1 (first contact with the healthcare system and linkage-to-care), M3 (linkage-to-care and initiation of ARV treatment), M6, M9 and M12 (medical follow-up and retention in care). Blood samples will be collected using Dried Blood Spot testing (DBS) at enrolment, M6 and M12. Furthermore, data will be collected about the characteristics of the healthcare centers around the artisanal gold mining sites (i.e. healthcare supply) and the costs of community-based HIV care.

The results will overcome the lack of epidemiological data about HIV in the informal gold mining zones, about the way in which PLWH are linked-to-care, and about the extent of the PLWH loss to follow-up. The results will also allow both testing the feasibility of the implementation of proximity community-based services for HIV care in the informal gold mining zones, and evaluating their contribution to retention of PLWH in care. The success of this project could allow extending the proposed strategy to other informal gold mining zones in Mali.

ELIGIBILITY:
Inclusion Criteria:

* To live and/or to work in the sites of Kofoulatiè or Diassa (Mali)
* To be diagnosed positive to HIV by ARCAD Santé PLUS (screening and enrolment tests positive)
* To be 18 years or older
* To speak one of the most common languages (Bambara, French or English) and to be able of providing informed consent

In addition, to be included in the intervention group, people living with HIV in the Kofoulatiè site must accept the community-based HIV care provided by ARCAD Santé PLUS

Exclusion Criteria:

* Women pregnant at the time of the HIV screening test by ARCAD Santé PLUS, or needing ultrasound to confirm pregnancy
* People with discordant screening and enrolment tests
* People inebriated or under the influence of drugs at enrolment
* Adults not able to understand and/or to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2020-11-29 (Actual); Primary Completion 2022-03-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Lost to follow-up rate 12 months after the HIV diagnosis | 12 months after HIV diagnosis (M12)
  It was defined on the basis of existing data: 1) lost to follow-up rate in HIV care at the national level in Mali (32% in 2019); 2) lost to follow-up rate in the HIV care of ARCAD Santé PLUS in urban areas (12% in 2019).
  The primary endpoint is : the lost to follow-up rate in the community-based HIV care 12 months after diagnosis is (at least) 20 percentage points lower than the lost to follow-up rate in the classic HIV care.

SECONDARY OUTCOMES:
Extent of the HIV epidemic in the artisanal gold-mining sites | At enrolment (M0)
  This outcome provides the prevalence of the HIV epidemic among people living/working in the artisanal gold-mining sites:
  number of HIV positive tests as percentage of the total number of people living/working in the sites
Comparing linkage-to-care and retention between classic and community-based HIV care | 1 month after HIV diagnosis (M1) and 12 months after HIV diagnosis (M12)
  For linkage-to-care:
  Percentage of people living with HIV starting a treatment 1 month and 3 months after diagnosis
  Percentage of people living with HIV with available blood tests (CD4 count, Viral load, etc) at the beginning of ARV treatment
  For retention in care:
  % of people living with HIV present for HIV care visits at 3, 6, 9 and 12 months after diagnosis
Comparing the impact of classic and community-based HIV care on virological succes, behavioral and psychosocial outcomes | From enrolment (M0) to 12 months after HIV diagnosis (M12)
  CD4 count and viral load at the time of diagnosis (M0) and its evolution 6 and 12 months later (M6 and M12)
  Self-perception of health status, sexual behavior indicators at M1 and evolution at M12: number of partners, number of sexual intercourses, etc.

OTHER OUTCOMES:
Material and human resources available for healthcare supply around gold-mining zones | From enrolment (M0) to 12 months after HIV diagnosis (M12)
  Description of the healthcare supply geographical distribution around the artisanal gold-mining zones included in the study;
  Description of the available human and material resources in the healthcare centers around the artisanal gold-mining zones included in the study
Working conditions of healthcare professionals involved in the classic HIV care | From enrolment (M0) to 12 months after HIV diagnosis (M12)
  Description of the socioeconomic and demographic characteristics of healthcare professionals in HIV care centers around the artisanal gold-mining zones included in the study;
  Number of working hours, number of medical visits, earnings, perceived health status, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sagaon Teyssier, PhD, Principal Investigator — UMR1252 SESSTIM (INSERM, IRD, Aix Marseille Université); Bintou Dembélé Keïta, MD, Principal Investigator — ARCAD Santé PLUS
Locations (4):
- Mali (4):
  - ARCAD Santé PLUS mobile care unit for community-based HIV care and study follow-up (Kofoulatiè, intervention site), Kofoulaté, Koulikoro
  - ARCAD Santé PLUS mobile care unit for recruitment of participants (Kofoulatiè, Intervention site), Kofoulaté, Koulikoro
  - ARCAD Santé PLUS mobile care unit for recruitment of participants (Diassa, control site), Diassa, Sikasso
  - Referral health center (CSRéf) Kolondieba, classic HIV care, Kolondiéba, Sikasso